CLINICAL TRIAL: NCT06458361
Title: Identification of Risk Factors and Construction of Prediction Model for Postoperative Intestinal Anastomotic Leakage in Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yang Shen, Vice-President, Chief Physician, Professor, Zhongda Hospital
Other Study IDs: 2024040145
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer
Keywords: Anastomotic Leakages; Risk Factors; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Anastomotic Leak | interventions — Aging; Body Mass Index; Marital Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anastomotic Leakage: Anastomotic Leakage in the first month after surgery
  Interventions: Procedure: Type of bowel resection, surgical complexity score, intraoperative blood loss, perioperative erythrocyte transfusion, type of anastomosis
- non-anastomotic Leakage: non-anastomotic Leakage in the first month after surgery
  Interventions: Procedure: Type of bowel resection, surgical complexity score, intraoperative blood loss, perioperative erythrocyte transfusion, type of anastomosis

INTERVENTIONS:
Procedure: Type of bowel resection, surgical complexity score, intraoperative blood loss, perioperative erythrocyte transfusion, type of anastomosis — Basic information about ovarian cancer patients and factors associated with preoperative, intraoperative and postoperative periods
  Other Names: Age, BMI, marital status, history of hypertension, history of diabetes mellitus

SUMMARY:
This study was a multicenter, retrospective cohort study. Although advancements in surgical techniques have mitigated the incidence of intestinal anastomotic fistula, complete avoidance remains elusive. Anastomotic leakage (AL) complications directly impinge on postoperative quality of life and pose life-threatening risks if inadequately managed. Given AL's adverse prognostic implications and the financial strain on patients' families, identifying its risk factors aids in perioperative risk assessment, enabling timely clinical decisions on interventions to enhance prognosis and curtail adverse outcomes and economic investments.

DETAILED DESCRIPTION:
Optimal cytoreduction, particularly in advanced cases, significantly extends 5-year survival compared to cases with residual disease exceeding 1 cm. Consequently, ultra-radical tumor cytoreduction procedures, commonly performed in advanced ovarian cancer, entail the excision of abdominopelvic tissues affected by the primary ovarian malignancy, including segments of the bowel, bladder, spleen, gallbladder, diaphragm, and other organs. Rectosigmoid resection (RSR) emerges as the predominant bowel resection, followed by colon and small bowel resections. Intestinal anastomosis post-RSR is indispensable for bowel reconstruction but bears a notable risk of postoperative anastomotic fistula (AL), a major complication. AL incidence rates fluctuate over time, reported between 8-14% in OC surgery patients undergoing RSR.

AL imposes considerable burdens, encompassing elevated hospital costs, prolonged stays, heightened rates of secondary admissions and surgeries, and mortality rates ranging from 3% to 21%. Furthermore, AL delays the commencement of adjuvant chemotherapy, detrimentally impacting overall survival and representing a significant consequence of colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with postoperative pathological diagnosis of primary ovarian, fallopian tube or peritoneal cancer
2. Patients undergoing tumour cytoreductive surgery combined with colorectal resection and stage I intestinal anastomosis
3. No history of other malignant tumours
4. Complete case data

Exclusion Criteria:

1. Previous combination of malignant tumours of other organs
2. Comorbidities with serious diseases related to other organs
3. Patients undergoing secondary tumour cytoreduction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients undergoing colorectal resection for patients with ovarian, fallopian tube and peritoneal cancer from January 2018 to June 2023 from multiple study centres were selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Risk Factors and a Prediction Model for Postoperative Intestinal Anastomotic Leakage in Ovarian Cancer | 1 month after surgery
  Risk Factors

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No